CLINICAL TRIAL: NCT03610815
Title: Community I-STAR Mozambique: Community Implementation of SBIRT Using Technology for Alcohol Use Reduction in Mozambique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Milton L. Wainberg, MD, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 7493
Record Dates: First submitted 2018-06-24; First posted 2018-08-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: mSBIRT - Mobile Screening, Brief Intervention, Referral to Treatment; SBIRT-CTS - Screening, Brief Intervention, Referral to Treatment Conventional Training and Supervision Strategy
Keywords: Alcohol; SBIRT; Mobile Technology; Implementation Science; Dissemination Research; Hybrid Effectiveness-Implementation Design
MeSH Terms: interventions — Mass Screening; Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation Hybrid 2 Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mSBIRT (Experimental): Mobile Screening, Brief Intervention, Referral to Treatment (mSBIRT)
  Interventions: Behavioral: Screening, Brief Intervention, Referral to Treatment
- SBIRT-CTS), (Active Comparator): Screening, Brief Intervention, Referral to Treatment Conventional Training and Supervision strategy
  Interventions: Behavioral: Screening, Brief Intervention, Referral to Treatment

INTERVENTIONS:
Behavioral: Screening, Brief Intervention, Referral to Treatment — Screening, Brief Intervention, Referral to Treatment
  Other Names: Motivational Interviewing

SUMMARY:
Hazardous drinking (HD) is a major public health burden worldwide with significant morbidity and mortality. To reduce HD, the World Health Organization (WHO) recommends using Screening, Brief Intervention, Referral to Treatment (SBIRT). Mobile health technology (mHealth), such as the mSBIRT app, is a promising tool for widespread cost-effective delivery of evidence-based HDS by community health workers (CHWs) because of its potential to increase fidelity, effectiveness, and sustainability. Community I-STAR Mozambique comprises three phases: 1) mSBIRT adaptation, 2) a cluster-randomized trial, and 3) scale-up of the most cost-effective intervention. Community I-STAR Mozambique will scale-up a cost effective, sustainable program and inform policy applicable to Mozambique and other LMICs.

DETAILED DESCRIPTION:
Hazardous drinking (HD) is a major public health burden worldwide with significant morbidity and mortality. The prevention and treatment gap associated with this global burden requires that efficacious interventions be scaled-up, leveraging existing platforms and participation of policy makers ready to apply and sustain evidence-informed policies over time. To reduce HD, the WHO recommends using Screening, Brief Intervention, Referral to Treatment (SBIRT) and the mental health Gap Action Programme guidelines (mhGAP). As low- and middle-income countries (LMIC) embrace SBIRT and mhGAP for community based HD services (HDS), a main scale-up challenge is ensuring effectiveness, fidelity, and sustainability of services. Mobile health technology (mHealth), such as the mSBIRT app, is a promising tool for widespread cost-effective delivery of evidence-based HDS by community health workers (CHWs) because of its potential to increase fidelity, effectiveness, and sustainability. The proposed project, Community I-STAR (Implementation of SBIRT using Technology for Alcohol use Reduction) Mozambique, will leverage the following existing Mozambique Ministry of Health (MoH) programs: (1) a task-shifting strategy training psychiatric technicians (PsyTs) to use the mhGAP; (2) the WHO-funded epilepsy community program delivered by CHWs; and (3) an mHealth program for malaria, pneumonia, and diarrhea (inSCALE - Innovations at Scale for Community Access and Lasting Effects). These currently operating programs set the stage for the use of mSBIRT by CHWs to deliver community HDS in Mozambique and generate policy for scale-up of government-funded community HDS harnessing existing human resources. Community I-STAR Mozambique comprises three phases: 1) mSBIRT adaptation, 2) a cluster-randomized trial, and 3) scale-up of the most cost-effective intervention. A formative phase to adapt mSBIRT to Mozambique's context/culture, will be followed by a 2-year, cluster-randomized, hybrid effectiveness-implementation type 2 trial in 12 districts: 6 districts randomized to receive mSBIRT and 6 to an SBIRT Conventional Training and Supervision strategy (SBIRT-CTS), with both arms delivered by CHWs. The arm showing higher cost-effectiveness in the 2-year trial will be scaled up to the other 6 districts for 12 "cross-over" months. Throughout the trial and the "cross-over" scale-up, qualitative and process data will complement quantitative assessments to examine implementation, sustainability, and scale-up. This approach redefines work roles without requiring new human resources, and it comports with the MoH's commitment to implementing HDS. Evidence-based practices (SBIRT) will a) build capacity for complete task-shifting of sustainable community-HDS practices; and b) use implementation tools to examine implementation and effectiveness of two SBIRT delivery strategies followed by evaluation of scale-up of the most cost-effective strategy. Community I-STAR Mozambique will scale-up a cost effective, sustainable program and inform policy applicable to Mozambique and other LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Community Health Workers working in the randomized clinics, Portuguese speakers

Exclusion Criteria:

* Other clinic staff from this clinics or other clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Implementation - Reach | From baseline to 6 months
  Number of individual who access care from among those who need care
Clinical Effectiveness - AUDIT | From baseline to 6 months
  Alcohol Use Disorders Identification Test

SECONDARY OUTCOMES:
Cost of Implementing New Strategies (COINS) | through study completion, an average of 2 years
  Measures cost of implementing interventions

CONTACTS AND LOCATIONS:
Overall Officials: Milton L Wainberg, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- MIHER: Mozambique Institute for Health Education and Research, Maputo, Cidade de Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Investigators will use the Global Mental Health Program at Columbia University (GMHP@CU) to make data available requiring acknowledgement of the the source of data and anonymity of research participants. Public codebooks and analysis protocols will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after study completion
Access Criteria: Described above in the plan description

REFERENCES:
- [Background] Morgenstern J, Irwin TW, Wainberg ML, Parsons JT, Muench F, Bux DA Jr, Kahler CW, Marcus S, Schulz-Heik J. A randomized controlled trial of goal choice interventions for alcohol use disorders among men who have sex with men. J Consult Clin Psychol. 2007 Feb;75(1):72-84. doi: 10.1037/0022-006X.75.1.72. PMID 17295566
- [Background] Irwin TW, Morgenstern J, Parsons JT, Wainberg M, Labouvie E. Alcohol and sexual HIV risk behavior among problem drinking men who have sex with men: An event level analysis of timeline followback data. AIDS Behav. 2006 May;10(3):299-307. doi: 10.1007/s10461-005-9045-7. PMID 16482407
- [Background] Elliott JC, Aharonovich E, O'Leary A, Wainberg M, Hasin DS. Drinking motives as prospective predictors of outcome in an intervention trial with heavily drinking HIV patients. Drug Alcohol Depend. 2014 Jan 1;134:290-295. doi: 10.1016/j.drugalcdep.2013.10.026. Epub 2013 Nov 5. PMID 24286967
- [Background] Elliott JC, Aharonovich E, O'Leary A, Wainberg M, Hasin DS. Drinking motives among HIV primary care patients. AIDS Behav. 2014 Jul;18(7):1315-23. doi: 10.1007/s10461-013-0644-4. PMID 24165984
- [Background] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593
- [Background] Aharonovich E, Hatzenbuehler ML, Johnston B, O'Leary A, Morgenstern J, Wainberg ML, Yao P, Helzer JE, Hasin DS. A low-cost, sustainable intervention for drinking reduction in the HIV primary care setting. AIDS Care. 2006 Aug;18(6):561-8. doi: 10.1080/09540120500264134. PMID 16831783
- [Background] Oquendo MA, Duarte C, Gouveia L, Mari JJ, Mello MF, Audet CM, Pinsky I, Vermund SH, Mocumbi AO, Wainberg ML. Building capacity for global mental health research: challenges to balancing clinical and research training. Lancet Psychiatry. 2018 Aug;5(8):612-613. doi: 10.1016/S2215-0366(18)30097-X. Epub 2018 Apr 5. No abstract available. PMID 29628365
- [Derived] Suleman A, Mootz JJ, Feliciano P, Nicholson T, O'Grady MA, Wall M, Mandell DS, Stockton M, Teodoro E, Anube A, Novela A, Mocumbi AO, Gouveia L, Wainberg ML. Scale-Up Study Protocol of the Implementation of a Mobile Health SBIRT Approach for Alcohol Use Reduction in Mozambique. Psychiatr Serv. 2021 Oct 1;72(10):1199-1208. doi: 10.1176/appi.ps.202000086. Epub 2021 Jun 15. PMID 34126774